CLINICAL TRIAL: NCT06185153
Title: Carbapenem Antibiotic Therapy for VIM Carbapenemase-Producing Enterobacteriaceae Infections - A Retrospective Cohort Study
Brief Title: Carbapenem Antibiotic Therapy for VIM Carbapenemase-Producing Enterobacteriaceae Infections
Acronym: CarbaVim
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8779
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Carbapenemase-Producing Enterobacteriaceae
Keywords: Carbapenemase; Enterobacteriaceae; VIM-producing strains

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Carbapenemase-producing Enterobacteriaceae (CPE) infections are emerging infections that pose a therapeutic challenge. These infections mainly occur in patients with prolonged hospitalization and repeated exposure to antibiotics. Certain strains, notably VIM-producing strains, may remain sensitive to carbapenems. CPE VIM strains are rare in France, but represent the main CPE strains in many countries. They are historically the main type of carbapenemases isolated at the Strasbourg University Hospital.

DETAILED DESCRIPTION:
The circulation of multi-antibiotic-resistant bacterial strains is significant at the Strasbourg University Hospital and the investigators wish to report their local experience in the use of carbapenems in infections with enterobacteria producing carbapenemase type VIM.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18)
* Treated at the HUS for a VIM-producing enterobacteria infection between 01/01/2011 and 11/30/2022
* Subjects who have not expressed their opposition to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Patient having expressed his opposition to the retrospective reuse of his data for scientific research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult patient (≥18) treated at the HUS for a VIM-producing enterobacteria infection between 01/01/2011 and 11/30/2022
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Mortality at 28 days | Mortality at 28 days after infection

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France